CLINICAL TRIAL: NCT02285855
Title: Tumor Mutation Status Will Predict Metabolic Response to Metformin in Non Small Cell Lung Cancer (NSCLC)
Brief Title: Metformin in Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0255; NCI-2015-00287 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non small cell lung cancer; Stereotactic body radiotherapy; SBRT; XRT; Radiation therapy; Metformin; Metformin ER; Placebo; Sugar pill; Lung adenocarcinoma; Genotypes; Genetic mutations
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Metformin; Sugars; Radiosurgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stereotactic body Radiotherapy (SBRT) + Metformin (Experimental): Participants randomized to Metformin treatment receive Metformin for 3 weeks prior to SBRT treatment and for 1 week during SBRT treatment. Metformin administered at a dose of 2000 mg by mouth in divided dose daily (500 mg am, 1000 mg noon, 500 mg pm). To reduce GI toxicity, participants start Metformin at 1000 mg daily in a divided dose (500mg am, 500 mg pm) for 1 week. SBRTdelivered per standard of care practice.
  Interventions: Drug: Metformin; Radiation: Stereotactic body Radiotherapy (SBRT)
- Stereotactic Body Radiotherapy (SBRT) + Placebo (Placebo Comparator): Participants randomized to placebo treatment 3 weeks prior to SBRT treatment and for 1 week during SBRT treatment. Placebo administered by mouth three times a day. SBRT delivered per standard of care practice.
  Interventions: Other: Placebo; Radiation: Stereotactic body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Metformin — Metformin treatment given at a dose of 2000 mg by mouth in divided dose daily (500 mg am, 1000 mg noon, 500 mg pm). To reduce GI toxicity, participants start Metformin at 1000 mg daily in a divided dose (500mg am, 500 mg pm) for 1 week.
  Other Names: Metformin ER
  Arms: Stereotactic body Radiotherapy (SBRT) + Metformin
Other: Placebo — Placebo treatment given 3 weeks prior to SBRT treatment and for 1 week during SBRT treatment. Placebo administered by mouth three times a day.
  Other Names: Sugar pill
  Arms: Stereotactic Body Radiotherapy (SBRT) + Placebo
Radiation: Stereotactic body Radiotherapy (SBRT) — SBRT delivered per standard of care practice as determined by participant's physician.
  Other Names: SBRT; XRT

SUMMARY:
The goal of this clinical research study is to learn if giving metformin in combination with radiation therapy is more effective than radiation therapy alone. In this study, participants will receive either metformin or a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

This is an investigational study. Metformin is FDA approved for the treatment of diabetes. Its use in this study to be given with radiation therapy to treat lung cancer is investigational. The study doctor can explain how the study drug is designed to work.

Up to 70 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic diagnosis of lung NSCLC or squamous cell carcinoma.
2. Patients are to be treated with hypofractionated RT.
3. Patient is not a surgical candidate due to medical comorbidities determined by a thoracic surgeon or patient refusal
4. Patient plans to receive treatment at MD Anderson
5. Patients must sign informed consent
6. Patient must have adequate renal function within 30 days prior to registration, defined as serum creatinine within normal institutional limits or creatinine clearance at least 60 ml/min

Exclusion Criteria:

1. Patient has: random glucose >200 mg/dl or is taking an oral hypoglycemic agent or insulin at the time of study entry
2. Patient has a history of lactic acidosis, chronic kidney disease or a creatinine >/= 1.2 mg/dl
3. Women who are pregnant or breast feeding, as treatment involves unforeseeable risks to the participant, embryo, fetus, or nursing infant
4. Patients with history of allergic reaction to metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G. Chun, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chun SG, Liao Z, Jeter MD, Chang JY, Lin SH, Komaki RU, Guerrero TM, Mayo RC, Korah BM, Koshy SM, Heymach JV, Koong AC, Skinner HD. Metabolic Responses to Metformin in Inoperable Early-stage Non-Small Cell Lung Cancer Treated With Stereotactic Radiotherapy: Results of a Randomized Phase II Clinical Trial. Am J Clin Oncol. 2020 Apr;43(4):231-235. doi: 10.1097/COC.0000000000000632. PMID 31990759
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 lung non-small cell lung cancer (NSCLC) patients were consented and randomized. Eligible criteria: pathologic diagnosis of AJCC Stage I-II, cT1-T2N0M0, can be treated with hypofractionated radiotherapy, not a surgical candidate, have adequate renal function within 30 days prior to registration, and plans to receive treatment at MDACC.
Pre-assignment Details: A total of 27 patients were consented to this study, but 9 patients withdrew consent prior to protocol medication or treatment. 18 patients randomized and treated under this protocol.
Groups:
- Metformin Arm: Patients randomized to metformin arm will receive 3 weeks of daily metformin (500 mg, am, 1000 mg, noon, 500 mg, pm) and then SBRT to a total dose of 50-70 Gy in 4-15 daily treatment fractions with metformin.
- Placebo Arm: Patients randomized to placebo treatment will receive 3 weeks of daily placebo and then SBRT to a total dose of 50-70 Gy in 4-15 daily treatment fractions with placebo.
Period: Overall Study
Arm/Group | Metformin Arm | Placebo Arm
Started | 16 | 2
Randomized | 16 | 2
Completed | 14 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 18 stage I non-small cell lung cancer (NSCLC) patients were consented and randomized. Metformin Arm 16 patients and Placebo Arm 2 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Arm | Placebo Arm | Total
Number analyzed (Participants) | 16 | 2 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 13 | 2 | 15
Age, Continuous [Median (Full Range); unit: Years] | 73.3 [52 to 84] | 69.3 [68 to 71] | 71.3 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 14 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 2 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 2 | 18
Total 15 patients completed treatment under the protocol and evaluable for data analysis. [Number; unit: Participants] — Three patients can not complete the treatment ( Metformin Arm in 2 and Placebo Arm in 1). There were 15 patients completed treatment. Randomized to placebo in 1 and to metformin in 14. American Joint Committee on Cancer [AJCC] 7th Ed: Stage IA: T1a, b N0 M0 Stage IB: T2a N0 M0 , T1a: primary tumor ≤2 cm, T1b: primary tumor >2-3 cm, T2a: primary tumor >3-5 cm, The earlier TNM staging, the better treatment outcome
  Participants
    (AJJC) Disease Stage 1A | 3 | 1 | 4
    (AJJC) Disease Stage 1B | 11 | 0 | 11
    (AJJC) Disease T Stage T1a | 2 | 1 | 3
    (AJJC) Disease T Stage T1b | 1 | 0 | 1
    (AJJC) Disease T Stage T2a | 11 | 0 | 11
    Tumor Histology Adenocarcinoma | 9 | 1 | 10
    Tumor Histology Squamous Cell Carcinoma | 4 | 0 | 4
    Tumor Histology Poorly differentiated carcinoma | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: RECIST and PERCIST Tumor Response
Description: The primary objective is the effect of metformin on response in NSCLC patients treated with hypofractionated RT. All patients will receive FDG-PET/CT scan at baseline (prior to metformin start), prior to RT and at 6 months (+/- 30 days) following RT. PET/CT imaging using [18F]-2-fluoro-2-deoxyglucose positron emission tomography (18F-FDG), using a standard approved radiopharmaceutical dose and administration selected by the nuclear medicine physician (120 min). Response will be determined at 6 months post-treatment via relative change from pre-treatment tumor by Response Evaluation Criteria in Solid Tumor (RECIST) by complete response (CR), partial response (PR) and stable disease (SD) and PET Response Criteria in Solid Tumors (PERCIST) by stable metabolic disease (SMD), progressive metabolic disease (PMD) and complete metabolic response(CMR).
Time Frame: From baseline (prior to metformin start) to Post-Radiotherapy (RT) Treatment, assessed up to 6 months
Population: Three participants did not complete the treatment ( Metformin Arm in 2 and Placebo Arm in 1). 15 participants randomized and completed ( Placebo Arm in 1 and Metformin Arm in 14). One participant died prior post treatment 6 months evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Arm | Placebo Arm
Number analyzed (Participants) | 14 | 1
Participants
  Mid-treatment RECIST tumor response (SD) | 14 | 1
  Post-treatment (6 mo.) RECIST tumor response(CR): number analyzed (Participants) | 13 | 1
  Post-treatment (6 mo.) RECIST tumor response(CR) | 7 | 1
  Post-treatment (6 mo.) RECIST tumor response(PR): number analyzed (Participants) | 13 | 1
  Post-treatment (6 mo.) RECIST tumor response(PR) | 3 | 0
  Post-treatment (6 mo.) RECIST tumor response(SD): number analyzed (Participants) | 13 | 1
  Post-treatment (6 mo.) RECIST tumor response(SD) | 3 | 0
  Mid-treamtment PERCIST tumor response: (SMD) | 6 | 1
  Mid-treamtment PERCIST tumor response: (PMD) | 6 | 0
  Mid-treamtment PERCIST tumor response: (PMR) | 2 | 0
  Post- treatment (6 mo.) PERCIST (CMR): number analyzed (Participants) | 13 | 1
  Post- treatment (6 mo.) PERCIST (CMR) | 9 | 1
  Post- treatment (6 mo.) PERCIST (PMD): number analyzed (Participants) | 13 | 1
  Post- treatment (6 mo.) PERCIST (PMD) | 1 | 0
  Post- treatment (6 mo.) PERCIST (PMR): number analyzed (Participants) | 13 | 1
  Post- treatment (6 mo.) PERCIST (PMR) | 3 | 0

ADVERSE EVENTS:
Time Frame: From the time of registration through study completion and follow up, assessed up to 6 months
Description: Adverse Events report based on Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE 4.0). All in the study patient encounter or treatment areas should have access to a copy of these criteria from the start of protocol treatment. Attributable to the protocol treatment (definitely, probably, or possibly related) should be reported as well.
Arm/Group | Metformin Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/1
Other Adverse Events (participants affected / at risk) | 0/14 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin Arm (N=14) | Placebo Arm (N=1)
Diarrhea (Gastrointestinal disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02285855/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02285855/SAP_001.pdf